CLINICAL TRIAL: NCT00626119
Title: In Vivo Breast Imaging by Vibro-acoustography
Brief Title: Vibro-Acoustography Imaging in Finding Breast Microcalcifications and Lesions in Women
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mostafa Fatemi, PhD, Mayo Clinic
Other Study IDs: 729-01-0; P30CA015083 (NIH); CDR0000583249 (Registry Identifier: NCI)
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control
- diseased

SUMMARY:
RATIONALE: New diagnostic procedures, such as vibro-acoustography imaging, may be an effective method of finding microcalcifications and lesions in the breast.

PURPOSE: This clinical trial is studying how well vibro-acoustography imaging works in finding breast microcalcifications and lesions in women.

DETAILED DESCRIPTION:
OBJECTIVES:

* To further develop a new method of in vivo imaging of the breast using vibro-acoustography (VA) imaging.
* To demonstrate and evaluate the capability of VA imaging in detecting microcalcifications and lesions inside the human breast.

OUTLINE: Participants undergo vibro-acoustography (VA) imaging of the breast using ultrasonography over 90 minutes. Participants may also undergo further imaging using clinical ultrasonography.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Healthy participant
  * Proven microcalcifications and/or lesions in the breast
* Hormone status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant or nursing
* No condition that does not allow proper use of study imaging devices

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with and without breast masses
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2001-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Further development of a new method of in vivo imaging of the breast using vibro-acoustography (VA) imaging | one day

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Fatemi, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States